CLINICAL TRIAL: NCT02487784
Title: Ridge Augmentation Comparing the Clinical and Histologic Healing of a Cancellous Block Allograft Versus Corticocancellous Particulate Allograft Mixed With Autogenous Bone Chips
Brief Title: Ridge Augmentation: Particulate v/s Block Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Henry Greenwell, Director of Graduate Periodontics, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15.0530
Record Dates: First submitted 2015-06-19; First posted 2015-07-01 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss | interventions — abacavir

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Particulate allograft + autogenous bone. (Experimental): In the test arm of the study the treatment will include a mix of MinerOss CorticoCancellous Particulate allograft + autogenous bone chips.
  Interventions: Procedure: Particulate allograft + autogenous bone chips
- Block allograft (Active Comparator): The positive control treatment will include a block allograft plus Mineross corticocancellous particulate allograft.
  Interventions: Procedure: Block allograft

INTERVENTIONS:
Procedure: Block allograft — A cancellous block allograft plus corticocancellous particulate allograft will be used as the positive control treatment.
  Other Names: Cancellous block allograft
  Arms: Block allograft
Procedure: Particulate allograft + autogenous bone chips — The test arm of this study will include a mix of particulate bone allograft and autogenous bone chips.
  Other Names: Particulate + ABC
  Arms: Particulate allograft + autogenous bone.

SUMMARY:
The primary aims of this study are to compare the clinical and histologic results of bone regeneration with a cancellous block allograft versus MinerOss Cortico cancellous particulate allograft mixed with autogenous bone chips after 4 months of healing. Titanium reinforced hd-PTFE (Cytoplast) membrane GBR will be used to cover the bone grafts.

Specific Aim 1: To compare the baseline to 4 month change in clinical ridge width and height.

Specific Aim 2: To compare the histologic percent of vital and nonvital bone and trabecular space at 4 months.

The primary outcome variable is the change in horizontal ridge width. The secondary outcomes are the change in ridge height and the percent histologic composition of the augmented site.

DETAILED DESCRIPTION:
30 patients will be treated using the principles of guided bone regeneration and ridge augmentation. 15 test patients will receive a corticocancellous particulate allograft mixed with autogenous bone chips. The positive control group of 15 patients will receive a cancellous block allograft. Both the groups will receive a hd-PTFE (Cytoplast) barrier membrane. An allograft can be defined as bone that can be obtained from a different individual of the same species (human donor bone) whereas a autograft can be defined as bone that can be obtained from the same individual. Following flap reflection, vertical measurements will be done using a acrylic occlusal stent and horizontal measurements will be done using a specially designed caliper. Approximately 4 months post surgery, a trephine core will be taken from the grafted site immediately prior to the implant placement and submitted for histologic processing. The last step in the study will be to obtain a trephine core (2.7 X 6mm). After the core is harvested a dental implant will be placed. Implant placement should be considered a post study treatment procedure. There is no intent to investigate implant placement outcome. Step serial sections will be taken from each longitudinally sectioned core. The sections will be stained with hematoxylin and eosin. Ten slides per patient will be prepared with at least 4 sections per slide. For each patient 6 of 10 slides will be assessed. The mean percentages of vital and non vital bone and trabecular space will be determined for each patient by using an American Optical Microscope at 150X with a 10 X10 ocular grid. Histologic preparation will result in destruction of the trephine cores. Means and standard deviations will be calculated for all parameters. A paired t-test will be used to evaluate the statistical significance of the differences between initial and final data. An unpaired t-test will be used to evaluate statistical differences between the test and control groups.

ELIGIBILITY:
Inclusion Criteria:

* At least a one tooth area with a ridge defect, treatment planned to receive a dental implant. The site must be bordered by at least one tooth.
* Healthy person that is at least 18 years old.
* Patient understands and signs an informed consent approved by the University of Louisville Human Studies Committee.

Exclusion Criteria:

* Patients with debilitating systemic diseases, diseases that significantly affect the periodontium, or psychological problems that would interfere with treatment.
* Previous head and neck radiation or chemotherapy within the previous 12 months.
* Patients with known allergy to any of the materials that will be used in the study.
* Smokers.
* Patients on oral bisphosphonates > 3 years or any IV bisphosphonates.
* Patients who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Horizontal ridge width changes | 4 months
  Site width (horizontal) changes by comparing the pre- to the 4 month post- augmentation dimensions of hard tissues.

SECONDARY OUTCOMES:
Vertical ridge height changes | 4 months
  Site height (vertical) changes by comparing the pre- to the 4 month post-augmentation dimensions of hard tissues.
Histologic composition of the graft | 4 months
  Histologic composition at 4 month post graft. (Histologic percent vital bone, nonvital bone and trabecular space.)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Greenwell, DMD, MSD, Principal Investigator — Director of Graduate Periodontics, School of Dentistry, University of Louisville.